CLINICAL TRIAL: NCT00405951
Title: A Phase I/II Study of Obatoclax Mesylate (GX15-070MS) Administered Every 3 Weeks in Combination With Docetaxel to Patients With Relapsed or Refractory Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Safety and Efficacy of Obatoclax Mesylate (GX15-070MS)in Combination With Docetaxel for the Treatment of Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gemin X (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEM010
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — obatoclax; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Obatoclax Mesylate + Docetaxel (Experimental): Obatoclax Mesylate 250mL in combination with Docetaxel
  Interventions: Drug: Obatoclax mesylate 250 ml; Drug: Docetaxel

INTERVENTIONS:
Drug: Obatoclax mesylate 250 ml
Drug: Docetaxel

SUMMARY:
Defects in the apoptotic process can lead to the onset of cancer by allowing cells to grow unchecked when an oncogneic signal is present. Obatoclax is designed to restore apoptosis through inhibition of the Bcl-2 family of proteins, thereby reinstating the natural process of cell death that is often inhibited in cancer cells.

This is a multi-center, open-label, Phase I/II study of obatoclax administered in combination with docetaxel in 3-week cycles to patients with relapsed or refractory Non-Small Cell Lung Cancer. Treatment may be administered on an outpatient basis. No investigation or commercial agents or therapies other than those described herein may be administered with the intent to treat the patient's malignancy. Supportive care measures including those directed at controlling symptoms resulting from Non-Small Cell Lung Cancer are allowed.

ELIGIBILITY:
Inclusion Criteria:

* Pathological confirmation of Non-Small Cell Lung Cancer (NSCLC)
* Must have been previously treated with a single platinum-based chemotherapy regimen and shown evidence of disease progression; no further limitations
* Must have normal organ function
* Must be willing to submit to blood sampling for planned PK and PD analysis
* Must have the ability to understand and willingness to sign a written informed consent form

Exclusion Criteria:

* No other agents or therapies administered with the intent to treat malignancy
* Patients with prior exposure to obatoclax or docetaxel
* Uncontrolled, intercurrent illness
* Pregnant women and women who are breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2006-10; Primary Completion 2008-11 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
RECIST criteria with at least one lesion equal to or greater than 2.0cm using conventional technique or equal to greater than 1.0cm with spiral comupted tomography (CT) scan in a single dimension | 18 months
  Determine the response rate to obatoclax in combination with docetaxel and characterize the safety profile.; Determine the steady-state pharmacokinetic parameters and pharmacodynamic response.

SECONDARY OUTCOMES:
Peripheral blood counts; Bone marrow aspirates and biopsies | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean Viallet, MD, Study Director — Gemin X Pharmaceuticals
Locations (7):
- United States (7):
  - Mayo Clinic College of Medicine, Scottsdale, Arizona
  - Tower Oncology, Beverly Hills, California
  - Georgetown University, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - University of Maryland, Baltimore, Maryland
  - MedStar Research Institute, Baltimore, Maryland
  - Arlington Cancer Center, Arlington, Texas